CLINICAL TRIAL: NCT06874881
Title: Effectiveness of Aquatic and Land Exercises on Chronic Nonspecific Low Back Pain: A Randomised Study
Brief Title: Aquatic and Land Exercises for Chronic Low Back Pain
Acronym: AquaLand-CLBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NARS01072024
Record Dates: First submitted 2025-03-07; First posted 2025-03-13 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-03

CONDITIONS: Chronic Low Back Pain (Non-specific, Uncomplicated)
Keywords: Chronic low back pain; Aquatic therapy; Hydrotherapy; Water-based exercise; Exercise intervention; Land Exercise; Quality of life; Rehabilitation research; Functional Disability
MeSH Terms: interventions — Hydrotherapy; Aquatic Therapy

STUDY DESIGN:
Intervention Model Description: Parallel-group, Randomized Controlled Trial (RCT) design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aquatic Exercise Group (Experimental): The aquatic exercise session is approximately 45-60 minutes, thrice a week, for twelve weeks, 36 sessions total. They are supervised by an experienced researcher who is a qualified Physiotherapist. The one-hour session generally includes a warm-up, the main exercise session, and a cool-down period. The exercises include balance and agility training, cardio exercises, flexibility, upper and lower limb stretching and strengthening exercises, trunk rotations, etc. Additionally, the group receives back care education involving guidelines and recommendations for adopting good posture, self-management, and active lifestyle advice each week of the intervention. Also, the participants are given a participant education handbook containing all the information and resources about LBP.
  Interventions: Other: Aquatic Exercises
- Land Exercise Group (Active Comparator): The land exercise group will follow the same structured protocol as the aquatic exercise group regarding duration, frequency, and intensity.
  Interventions: Other: Land Exercises

INTERVENTIONS:
Other: Aquatic Exercises — The aquatic exercise intervention consists of structured, supervised, water-based exercises designed and delivered by an experienced physiotherapist specifically for individuals with chronic low back pain. Sessions are conducted in a temperature-controlled swimming pool with proper warm-up and cool-down. The intervention follows a progressive intensity approach with easy, medium, and hard approaches.
  Other Names: Aquatic Physical Therapy; Hydrotherapy; Water-Based Exercises; Aquatic Therapy; Pool-Based Rehabilitation; Aquatic Physiotherapy; Aquatic Rehabilitation; Therapeutic Water Exercise
  Arms: Aquatic Exercise Group
Other: Land Exercises — The land-based exercise intervention mirrors the aquatic exercise protocol regarding exercise type, duration, frequency, and progression but is performed on land.
  Other Names: Land-Based Exercise Therapy; Physiotherapy-Based Exercise; Musculoskeletal Rehabilitation Program; Therapeutic Exercise Routine
  Arms: Land Exercise Group

SUMMARY:
This study aims to learn about the effects of aquatic and land exercises on managing chronic low back pain in adults aged 18-65. The participants engage in a 12-week supervised land and water-based exercise program.

The main questions this study aims to answer are:

* How effective are aquatic exercises on low back pain, functional disability, Kinesiophobia, sleep quality, and overall quality of life?
* Is aquatic therapy more effective than land exercises for treating LBP or vice versa?

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65
* Both Genders
* Literate in the English language to understand instructions/ to complete a self-report questionnaire.
* Having non-specific Chronic low back pain (≥12 weeks)
* Patient willingness to be a part of any randomly selected treatment groups.

Exclusion Criteria:

* Pregnant Females
* If they had low back pain as the result of diagnosis of severe osteoporosis, spinal bone disorders such as spondylosis and spondylolisthesis, fractures, lumbar spine stenosis, lower limb joint replacement surgery, hip orthosis, ankylosing spondylitis, rheumatoid arthritis, infective or inflammatory disease, compression of the radial nerve, meningitis, arthrosis, lumbar region tumours, Leg length discrepancy, previous back surgery.
* Uncontrolled hypertension, Severe postural hypotension, any heart disease like Left heart failure or exercise-induced angina. Medical illnesses without a medical managing plan in place, e.g., uncontrolled epilepsy, diabetes mellitus. Neurologic deficit, open wounds, current or recurrent radiation treatment.
* Patients with severe depression and psychosis
* People who are already participating in an individually-prescribed exercise programme for LBP.

Aquatic exercises /Pool specific:

* Individuals with hydrophobia/ water-related anxiety, or inability to adapt to an aquatic environment.
* Allergy to chlorine, Severe limiting airway disease
* Faecal or urinary incontinence, diarrhoea, and vomiting.
* Weight more than the emergency evacuation manual handling risk assessment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2025-03-06 (Actual); Primary Completion 2025-11-28 (Actual); Study Completion 2025-11-28 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | Baseline before the intervention/pre-testing, at the 8th week of the intervention, within a week after the last training session, and three months after the end of the training (Follow-up period).
  Pain intensity is measured by the Numerical Pain Rating Scale where the participants will report their pain as 0 (no pain) and 10(worst imaginable pain).
Functional Disability | Baseline before the intervention/pre-testing, at the 8th week of the intervention, within a week after the last training session, and three months after the end of the training (Follow-up period).
  Functional disability is assessed by the Roland-Morris Disability Questionnaire, a 24-item self-reported measure evaluating the impact of low back pain on daily activities.

SECONDARY OUTCOMES:
Health-Related Quality of Life | Baseline before the intervention/pre-testing, at the 8th week of the intervention, within a week after the last training session, and three months after the end of the training (Follow-up period).
  Quality of Life is assessed by the Short-Form Health Survey 36, a validated questionnaire measuring the eight physical and mental health domains.
Sleep Quality | Baseline before the intervention/pre-testing, at the 8th week of the intervention, within a week after the last training session, and three months after the end of the training (Follow-up period).
  The Pittsburgh Sleep Quality Index measures the sleep quality, its scores measured from 0-21, with higher scores indicating poor sleep quality.
Kinesiophobia (Fear of Movement-Related to Pain) | Baseline before the intervention/pre-testing, at the 8th week of the intervention, within a week after the last training session, and three months after the end of the training (Follow-up period).
  Kinesiophobia is measured with the Tampa Scale of Kinesiophobia, a 17-item questionnaire designed to measure the fear associated with the chronic pain and movement.
Dynamic Balace Performance | Baseline before the intervention/pre-testing, at the 8th week of the intervention, within a week after the last training session, and three months after the end of the training (Follow-up period).
  The Y balance test measures dynamic balance by measuring stability while reaching in three directions: anterior, posteromedial, and posterolateral.
Hamstring Flexibility | Baseline before the intervention/pre-testing, at the 8th week of the intervention, within a week after the last training session, and three months after the end of the training (Follow-up period).
  The active knee extension test is a clinical measure of the hamstring flexibility.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Leonard building, The University of Edinburgh, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No